CLINICAL TRIAL: NCT05879848
Title: Synchronization of a VR Scenario to Uterine Contractions for Labor Pain Management: Development Study and Randomized Controlled Trial
Brief Title: VR Scenario for Labor Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Laura Sarno, Principal Investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FEDIIU485/20
Record Dates: First submitted 2023-04-02; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental analgesic treatment (VR) (Experimental): Achieved active labor and regular contractions (>= 4 contractions in 10 minutes), patients are given the virtual reality scenario synchronized with the uterine contractions , and no other alternative analgesia is provided, except for the midwife's support.
  Interventions: Other: VR
- Standard Care (non-VR) (No Intervention): Patients in active labour. undergo standard care (only midwife's support, no analgesia)

INTERVENTIONS:
Other: VR — virtual reality scenario synchronized with the uterine contractions
  Arms: Experimental analgesic treatment (VR)

SUMMARY:
The present study aims to evaluate Virtual Reality analgesic interventions for active labor with biofeedback-based Virtual Reality technologies synchronized to uterine activity. The investigators developed a Virtual Reality system modeled on uterine contractions by connection to a cardiotocographic equipment. The present study, based on a multidisciplinary approach, comprised the following phases: 1)development of hardware and software components; 2) design of the Reality scenario through a qualitative focus group discussion study; 3) clinical trial on a sample of 53 cases and 53 controls during active labor.

DETAILED DESCRIPTION:
Labor is described as one of the most painful events women can experience throughout their lives. A severe labor pain can have long lasting effects, as a severe labor can affect breastfeeding and is associated with an increased risk of postpartum depression. The current gold standard for labor pain management is pharmacological pain management techniques. However, their application is still flawed by its invasiveness, potential collateral effects, and financial. Consequently,researchers have investigated the role of complementary and alternative medicine in reducing labor pain like Virtual reality, that is a technology that allows users to immerse themselves in a three dimensional computer-generated scenario. At present, many studies have tested Virtual Reality interventions for the pain management of chemotherapy infusions, acute burn injuries, cancer-related and, recently, labor pain. The present study aimed to develop a biofeedback-implemented Virtual Reality scenario through algorithm-based cardiotocographic pattern processing that can effectively reduce labor anxiety and fear of labor and generally induce a positive emotional state during use.

Materials and Methods:

The study relied on a multidisciplinary team involving a psychologist, a gynecologist, three software engineers, a midwife, and a psychiatry resident to develop a biofeedback implemented Virtual Reality system. The interdisciplinary team conducted brainstorming sessions and discussed the development of the new system in light of the previous literature on the topic.

System development: the functioning of the developed system and its components. Hardware components: 1) Fetal monitor: Philips Avalon 2) Philips Avalon Fetal and Maternal Cableless Pod 3)Oculus Quest 2 Virtual Reality head-mounted display 4) Windows. Software components: 1) Medicollector SERVICE 2) Steam Virtual Reality 2.0. The system hardware architecture involves using the Meta Quest 2 head mounted display to immerse patients in a relaxing environment. Since the rendering of the virtual environment is performed on a computer, the investigators realize a more complex environment than what would have been possible by exploiting the computing capacity of the Head Mounted Display exclusively. However, in the system architecture, using a computer is due to two main reasons: i) to enable obstetricians to monitor the activities of laboring women and ii) to acquire physiological data from the cardiotocograph bonded to the patient. On this last one, the computer is physically connected to the cardiotocograph. Specifically, a Philips fetal monitor was used. The monitor is connected to the computer via a network cable and an adapter. The system prototype was developed using Unity 2019.4.14 and Steam Virtual Reality 2.0. Unity, one of the most popular cross-platform graphics engines for developing Virtual Reality applications, was used to create the virtual environment. The Steam Virtual Reality tool simplifies experiencing the Virtual Reality environment on the chosen Head Mounted Display. The fetal monitor data acquisition relies on the Medicollector software, executed on the computer, and the final application responsible for rendering the virtual environment and transmitting to the Head Mounted Display. Medicollector provides to access cardiotocography data, which can be used to access the fetal heart rate and uterine contractions for adapting the scenario each time a peak in the uterine contractions is detected.

Qualitative focus group discussion study: The scenario design resulted from a series of focus group sessions moderated by the psychologist of the multidisciplinary team. The second author was an observer attending the meetings and collecting notes. The volunteers were selected from women who had given birth at University Hospital "Federico II" of Naples. A total of 12 mothers were recruited and randomly assigned to three focus groups, each consisting of four mothers. After informed consent was obtained, the date and time of the meetings were arranged. Discussions took place between March and April 2021. The three focus groups lasted 89, 92, and 97 minutes and involved a semi-structured discussion divided into two parts. In the first part of the sessions, women were invited to discuss their childbirth experiences, their pain, and what helped them endure the contractions. In the second phase, after explaining the developed system and the purpose of the designed experimental intervention, women were invited to discuss how participants would imagine a virtual scenario that could have helped them relax and better stand the labor pain. Developed Virtual Reality scenario: The developed scenario involves a tropical beach lined with palm trees, surrounded by green mountains, and bathed by a calm sea. In the subject's immediate surroundings, an interactive virtual element was placed: a drum that could be played through the use of controllers. In addition, the scenario reproduced elements present in the actual labor room: the patient's bed and a cardiotocograph. The patient's bed position in the system reflected that of the real bed in the labor room, so users could reach the bed while wearing the Head Mounted Display. The cardiotocograph monitor was introduced into the environment so that patients could visually access the clinical parameters acquired by the cardiotocograph. During contractions, a flock of storks can be seen in the distance flying toward the subject's point of view. These have been placed in the environment with a twofold purpose: i) as a propitiatory message and ii) as a distracting element adaptive to the intensity of the detected uterine contractions. The adaptive system module displays the flock of storks in the virtual environment after detecting an incoming peak value of uterine contraction. Furthermore, in the scenario realized, when the storks are in flight, the storks can be attracted to the user's position by repeatedly playing the drum. If deemed appropriate or desired by the user, this element could also be activated manually by the medical and obstetrical staff via the computer keyboard. Intervention: Subjects randomly assigned to the intervention group were provided a Virtual Reality headset. Once active labor and pain intensity of regular contractions of 4/10 is reached, the virtual reality scenario synchronized to the uterine contractions is administered. During the procedure, no alternative analgesia methods are provided beside the continuous physical presence and vocal support of obstetric personnel. Immediately before and after using the headset, patients fill out the required questionnaires and scales.

ELIGIBILITY:
Inclusion Criteria:

* Single term pregnancy;
* Full term physiological pregnancy;
* Active phase of labor;
* Spontaneous labor;
* Nulliparous between 37 and 42 weeks of gestation with cephalic presentation;
* Maternal age between 18 and 45 years.

Exclusion Criteria:

* Twin pregnancy;
* Preterm labor;
* Preterm rupture of amnio membranes;
* Fetal abnormalities;
* Intrauterine growth restriction;
* Post-term pregnancy;
* Women with impaired consciousness, seriously ill, mentally disabled;
* Women under the age of 18 or over the age of 45;
* Women with visual and/or auditory impairments;
* Women prone to seizures;
* Women with a predisposition to motion sickness;
* Refusal to sign informed consent;
* Previous cesarean section.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Subjective pain | 1 year
  numerical rating scale for pain

SECONDARY OUTCOMES:
NAUSEA | 1 year
  numerical rating scale for nausea
Objective pain via wristband | 1 year
  heart rate measurement
incidence of episiotomy and lacerations | 1 year
  incidence of episiotomy and lacerations
epidural anesthesia | 1 year
  incidence of epidural anesthesia
incidence of operative delivery | 1 year
  incidence of use of vacuum extractor
neonatal outcome | 1 year
  APGAR score at 5 and 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: No